CLINICAL TRIAL: NCT04824495
Title: Evaluation of Inflammatory Cytokines During COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniela Gompelmann, Prof. Dr. med., University of Vienna
Other Study IDs: Version 1.1, 31.12.2021
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute COVID-19
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood samples at different timepoints during SARS-CoV2 infection

SUMMARY:
The aim of this study is to evaluate pro-inflammatory cytokines as well as microvesicles during the course of SARS-CoV2 infection in the context of clinical parameters.

DETAILED DESCRIPTION:
In this prospective trial, 100 patients with an acute SARS-CoV2 infection are enrolled. After confirmation of COVID-19, blood samples are taken for evaluation of various inflammatory cyokines and microvesicles at day 1, 5, 9 and 13 during hospitalisation and are interpreted in the context of clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmation of acute SARS-CoV2 infection
* Ability to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed acute SARS-CoV2 infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine level in context with clinical parameters | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gompelmann, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antoniewicz L, Melnikov G, Lyytinen G, Blomberg A, Bosson JA, Hedman L, Mobarrez F, Lundback M. Vascular Stress Markers Following Inhalation of Heated Tobacco Products: A Study on Extracellular Vesicles. Cardiovasc Toxicol. 2025 Jan;25(1):1-8. doi: 10.1007/s12012-024-09934-6. Epub 2024 Oct 29. PMID 39472409